CLINICAL TRIAL: NCT00291863
Title: Simvastatin Effect on Endothelium Dependent Venodilation in Chronic Renal Failure Patients Treated by Peritoneal Dialysis
Brief Title: Simvastatin Effect on End Stage Renal Failure Patients Treated by Peritoneal Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0089/04
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2006-02

CONDITIONS: Renal Failure, End Stage; Peritoneal Dialysis
Keywords: end stage renal failure; peritoneal dialysis; simvastatin; endothelium; vasodilation
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Aneurysm | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
This study will analyse the effect of simvastatin on endothelium dependent venodilation in chronic renal failure patients treated by peritoneal dialysis. The hypothesis is that patients will have a greater endothelium dependent venodilation after four months of simvastatin use.

DETAILED DESCRIPTION:
This study will analyse the effect of simvastatin on endothelium dependent venodilation in chronic renal failure patients treated by peritoneal dialysis. The hypothesis is that patients will have a greater endothelium dependent venodilation after four months of simvastatin use.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal failure
* peritoneal dialysis
* LDL cholesterol > 100mg/dL
* > 18 years and < 80 years

Exclusion Criteria:

* using statin or nitrate
* liver disease
* diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-02; Study Completion 2006-02

PRIMARY OUTCOMES:
endothelial venodilation

SECONDARY OUTCOMES:
Inflammation markers (C-reactive protein, IL-6, TNF)
Lipoproteins
Oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Maristela Bohlke, master, Principal Investigator — Federal University of São Paulo
Locations (1):
- São Lucas Hospital, Porto Alegre, Rio Grande do Sul, Brazil